CLINICAL TRIAL: NCT00328211
Title: Intralumenal Effects on Cholesterol Absorption/Synthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: DK68463; R01DK068463 (NIH)
Record Dates: First submitted 2006-05-18; First posted 2006-05-19 (Estimated); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: Healthy
MeSH Terms: interventions — Bile Acids and Salts; Sphingomyelins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bile Acid (Experimental): To assess the role of bile acid pool size changes on cholesterol absorption, synthesis and intralumenal cholesterol solubilization.
  Interventions: Dietary Supplement: Bile Acids (Cholic, Ursodeoxycholic, Chenodeoxycholic)
- Cholesterol Absorption (Experimental): To determine whether cholesterol absorption, synthesis and solubilization will be significantly altered by changes in phospholipid content, specifically sphingolipids and phosphatidylcholine in the intestinal lumen.
  Interventions: Dietary Supplement: Sphingomyelin
- Intralumenal (Experimental): To assess intralumenal solubilization and absorption of biliary and dietary cholesterol.
  Interventions: Dietary Supplement: Bile Acids (Cholic, Ursodeoxycholic, Chenodeoxycholic); Other: C13 Stable isotope of Cholesterol

INTERVENTIONS:
Dietary Supplement: Bile Acids (Cholic, Ursodeoxycholic, Chenodeoxycholic) — 15 mg/kg/day for 18 days
  Arms: Bile Acid; Intralumenal
Dietary Supplement: Sphingomyelin — 1000mg/day for 19 days
  Arms: Cholesterol Absorption
Other: C13 Stable isotope of Cholesterol — Food provided for 3 days and one time dose of 113mg of C13 Cholesterol.
  Arms: Intralumenal

SUMMARY:
The overall goal of this study is to better understand how cholesterol is absorbed and utilized in the body(metabolism) and how serum cholesterol affects the development of hardening of the arteries (atherosclerosis). The purpose of aim 1 is to assess the role of the amount of different bile acids in the intestine and how they affect the absorption, synthesis and digestion of cholesterol. The effect that these bile acids have on how fast the gall bladder empties and the release of a hormone in the blood after a meal will also be studied. The purpose of aim 2 is to assess the role of phospholipid (a fat containing the element phosphorus) in the intestine and how it affects the absorption, synthesis and digestion of cholesterol in normal people and in people with a genetic condition (mdr3 deficiency)that affects phospholipid and bile acid metabolism. The purpose of aim 3 is to assess the role of a material that acts like a detergent called Pluronic F-68 which is known to block the absorption of cholesterol. The purpose of aim 4 is to determine if the cholesterol from food and the cholesterol made by the body are digested and absorbed differently.

DETAILED DESCRIPTION:
Cholesterol absorption plays a key role in cholesterol homeostasis and understanding the lumenal events that play key roles in absorption remain poorly understood. The aims of the present study are fourfold: 1) To determine whether previously observed effects on cholesterol absorption during bile acid feeding are related to changes in pool size and intestinal transit or meal stimulated gall bladder emptying or plasma cholecystokinin levels. 2) To determine the effect of dietary sphingomyelin on cholesterol absorption, micellar solubilization and synthesis in normal adults and to assess the effects of intralumenal cholesterol solubilization, absorption and synthesis in adults with heterozygous mdr 3 deficiency (a defect leading to low biliary phospholipid content). 3) To determine the mechanism of action of a non-ionic detergent, Pluronic F-68, by evaluating its effect on cholesterol solubilization and distribution between micelles and vesicles, on cholesterol absorption and synthesis. 4) To evaluate the intralumenal solubilization and distribution within micelles and vesicles of biliary compared to dietary cholesterol in humans and assess the impact of ezetimibe treatment on absorption of endogenous or exogenous cholesterol by assessing absorption of human contents in the biliary diverted, rat lymph fistula model. For each of these aims, subjects will be studied while consuming well-controlled diets as outpatients with a combination of human and animal techniques. Techniques employed for human studies will include state-of-the art techniques utilizing stable isotopes and isotope ratio mass spectrometry, gas chromatography. Translational studies in animals will be used including novel techniques to measure fat absorption as well as the use of the lymph fistula rat model for assessment of lipid absorption and hamsters for assessment of bile acid and sterol synthesis. Integration of animal/human techniques will provide tools to characterize the role of modifications of the intralumenal environment on cholesterol solubilization and human cholesterol absorption and synthesis.

ELIGIBILITY:
Inclusion Criteria:

* Serum Total Cholesterol <200 mg/dl, LDL-Cholesterol <120 mg/dl
* Apo E-3/3, Apo A IV-1/1 genotypes

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus, other gastrointestinal, liver, kidney or heart disease
* Allergy to soy products

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2005-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The primary outcomes for this study are to better understand the molecular and cellular mechanisms of cholesterol metabolism and absorption. | 5 yrs

CONTACTS AND LOCATIONS:
Overall Officials: James E. Heubi, M.D., Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (1):
- Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yao L, Heubi JE, Buckley DD, Fierra H, Setchell KD, Granholm NA, Tso P, Hui DY, Woollett LA. Separation of micelles and vesicles within lumenal aspirates from healthy humans: solubilization of cholesterol after a meal. J Lipid Res. 2002 Apr;43(4):654-60. PMID 11907149
- [Background] Woollett LA, Buckley DD, Yao L, Jones PJ, Granholm NA, Tolley EA, Heubi JE. Effect of ursodeoxycholic acid on cholesterol absorption and metabolism in humans. J Lipid Res. 2003 May;44(5):935-42. doi: 10.1194/jlr.M200478-JLR200. Epub 2003 Mar 1. PMID 12611908
- [Background] Woollett LA, Buckley DD, Yao L, Jones PJ, Granholm NA, Tolley EA, Tso P, Heubi JE. Cholic acid supplementation enhances cholesterol absorption in humans. Gastroenterology. 2004 Mar;126(3):724-31. doi: 10.1053/j.gastro.2003.11.058. PMID 14988826
- [Background] Woollett LA, Wang Y, Buckley DD, Yao L, Chin S, Granholm N, Jones PJ, Setchell KD, Tso P, Heubi JE. Micellar solubilisation of cholesterol is essential for absorption in humans. Gut. 2006 Feb;55(2):197-204. doi: 10.1136/gut.2005.069906. PMID 16407385
- [Background] Ramprasath VR, Jones PJ, Buckley DD, Woollett LA, Heubi JE. Effect of dietary sphingomyelin on absorption and fractional synthetic rate of cholesterol and serum lipid profile in humans. Lipids Health Dis. 2013 Aug 19;12:125. doi: 10.1186/1476-511X-12-125. PMID 23958473